CLINICAL TRIAL: NCT06850402
Title: Evaluation of a Novel Optical Microscope With a Deep Depth of Field (DeepDOF) to Provide Histologic-quality Images on Cervical Biopsies and Loop Electrosurgical Excision Procedure (LEEP) Specimens at the Point-of-care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-2034; NCI-2025-01257 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-02-17; First posted 2025-02-27 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer; HIV
Keywords: HPV DNA Testing
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- DeepDOF Images (Experimental): Participants will be approached by a trained research assistant. After informed consent is obtained, each participant will collect two cervical swabs (self-collected and/or provider-collected) as an optional procedure and stored for future research. VIA and/or colposcopy will be performed per standard of care. Cervical biopsy(ies) and/or LEEP will be performed per standard of care. The specimens will be imaged immediately using DeeDOF at the point of care and then submitted for standard histopathologic analysis as shown in Figure 1.
  Interventions: Device: DeepDOF Images

INTERVENTIONS:
Device: DeepDOF Images — Women referred for consultation for cervical biopsy(ies) and/or LEEP will be recruited into the experimental group of the study.

SUMMARY:
All patients will be enrolled in Mozambique and Brazil. They will provide informed consent to use their cervical biopsy and/or LEEP specimens for imaging with DeepDOF prior to sending for standard of care processing and interpretation.

DETAILED DESCRIPTION:
Primary Objectives:

1. Evaluate the diagnostic performance of the DeepDOF digital histopathology platform compared with standard histopathology in cervical biopsies and/or LEEP specimens.
2. Compare performance characteristics between WLWH and HIV-negative women.

Secondary Objectives:

1. Evaluate the ability of pathologists to provide a diagnostic evaluation of cervical biopsies and LEEP margins using digital DeepDOF images.
2. Develop DeepDOF algorithms for automated diagnostic evaluation of cervical biopsies and LEEP margins.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 25 - 49 years
2. women undergoing cervical biopsy and/or LEEP
3. Women who are not pregnant and with a negative pregnancy test (within 3 days of enrollment)
4. Willing and capable of providing informed consent

Exclusion Criteria:

1. Women under 25 or over 49 years of age
2. Women not undergoing cervical biopsy or LEEP
3. Women who are pregnant

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 400 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary Out Measures | through study completion, an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Schmeler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org